CLINICAL TRIAL: NCT03657199
Title: Early Silent Graft Failure in Off-pump Coronary Artery Bypass Grafting: A Computed Tomography Analysis
Status: Completed | Type: Observational
Sponsor: Triemli Hospital (Other)
Responsible Party: Principal Investigator, Alicja Zientara, resident for cardiac surgery, Triemli Hospital
Other Study IDs: KEK-ID 2017-02315
Record Dates: First submitted 2018-08-30; First posted 2018-09-04 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Coronary Artery Disease; Bypass Complication; Graft Failure
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bypass graft failure: Patients with at least one detected graft failure after routine cardiac computed tomography before discharge
  Interventions: Diagnostic Test: Cardiac computed tomography
- No bypass graft failure: Patients without occluded bypass grafts after routine cardiac computed tomography before discharge
  Interventions: Diagnostic Test: Cardiac computed tomography

INTERVENTIONS:
Diagnostic Test: Cardiac computed tomography — Routine computed tomography of the heart before discharge

SUMMARY:
Aortocoronary bypass surgery is one of the most common operations in the western world. The goal of the surgeon is to perform a complete revascularization of the coronary arteries with the best, available bypass material.

Aortocoronary bypass surgery can be performed with (on-pump) or without (off-pump) the heart lung machine. If the operation is performed without the heart lung machine, the heart is continuously beating while the surgeon sews the bypass to the diseased coronary artery. In randomized trials, the benefits of the off-pump technique in the hands of experienced surgeons in terms of shorter operating times, less transfusions and less pulmonary and renal complications were proven. A criticism of the off-pump technique is the reduced number of distal anastomoses, which means that fewer coronary arteries may be connected with bypass grafts because of the technically sophisticated situation. A worse quality of the connection (anastomosis) between coronary artery and bypass is often discussed, leading to a bypass occlusion already in the early stage after surgery resulting in more re-interventions on the coronary vessels. So-called silent bypass failure without clinical correlation has been examined in three relevant studies including both, the on- and the off-pump technique, with inhomogenous results. In addition to the technique, other parameters such as the degree of narrowing (stenosis) of the diseased coronary artery and collateralization of a closed coronary artery may play a role in early occlusion.

All bypass patients after off-pump surgery receive routinely a computed tomographic examination of the heart. With this method, silent bypass occlusions without clinical correlation, i.e. cardiac infarction, elevated cardiac laboratory parameters or ECG changes, can be detected easily. In case of an occlusion of a relevant bypass, an intervention before discharge can be planned and performed.

We would like to investigate the occlusion rate of this retrospective patient cohort after off-pump surgery and the potential risk factors, that may influence on early graft failure. We hypothesize, that early graft failure depends not only on the choice of the graft material, but also on the local grade of coronary stenosis, the collateralisation of occluded coronary vessels and the intraoperative flow results, as well as on the region of the target vessel.

ELIGIBILITY:
Inclusion Criteria:

* patients after off-pump coronary artery bypass grafting
* postoperative computed tomography for the evaluation of the bypass patency before discharge

Exclusion Criteria:

* Operation with a heart-lung machine
* Combined interventions
* Postoperative emergency coronary angiography
* There is a documented rejection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients after off-pump coronary artery bypass grafting from January 2017 till April 2018, who received a postoperative computed tomography for the evaluation of the bypass patency before discharge
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Early postoperative graft failure | first week after aortocoronary bypass grafting
  Assessment of graft failure by computed tomography in all patients after isolated off-pump surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alicja Zientara, Dr, Principal Investigator — Triemli Hospital Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zientara A, Rings L, Bruijnen H, Dzemali O, Odavic D, Haussler A, Gruszczynski M, Genoni M. Early silent graft failure in off-pump coronary artery bypass grafting: a computed tomography analysisdagger. Eur J Cardiothorac Surg. 2019 Nov 1;56(5):919-925. doi: 10.1093/ejcts/ezz112. PMID 31006005